CLINICAL TRIAL: NCT03067857
Title: Autologous Purified Bone-Marrow-Derived Stem Cell Therapy for Motor Neuron Disease
Brief Title: Autologous Bone Marrow-Derived Stem Cell Therapy for Motor Neuron Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-MND1
Record Dates: First submitted 2017-02-25; First posted 2017-03-01 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Progressive Muscular Atrophy; Progressive Bulbar Palsies
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal; Bulbar Palsy, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cells (Experimental): Intravenous and Intrathecal thecal transplantation via interventional radiology of purified autologous bone-marrow derived specific stem cell populations.
  Interventions: Biological: Stem Cells

INTERVENTIONS:
Biological: Stem Cells — Autologous bone marrow-derived stem cell populations injected via the intravenous and intrathecal routes.

SUMMARY:
Herein, the investigators study the safety and efficacy of transplanting purified autologous bone marrow-derived stem cells transplanted via the intrathecal route by interventional radiology and the intravenous route.

DETAILED DESCRIPTION:
A motor neuron disease (MND) is any of several neurological disorders that selectively affect motor neurons, the cells that control voluntary muscles of the body. They include amyotrophic lateral sclerosis (ALS), primary lateral sclerosis (PLS), progressive muscular atrophy (PMA), progressive bulbar palsy (PBP) and pseudobulbar palsy; spinal muscular atrophies are also sometimes included in the group.They are neurodegenerative diseases that cause increasing disability and eventually, death.

In spite of intensive research, motor neuron diseases (MNDs) are still incurable. Some of the key factors in this failure to find a cure have been the lack of human cell-based disease models for molecular analysis and drug screening and the difficulty of obtaining homogeneous populations of specific cell types for clinical applications. Stem cell biology has the potential to transform our understanding of disease processes and to revolutionize our approach to develop novel therapies for MNDs.

In this study, the investigators suggest a protocol for the treatment of MND by transplantation of purified autologous bone marrow-derived stem cells via the intrathecal and intravenous route.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 24-20 years old
* Patients with the diagnosis of definite Motor Neuron Disease

Exclusion Criteria:

* HIV/HBV/HCV
* Malignancies
* Bleeding
* Pneumonia
* Renal failure
* liver dysfunction
* Severe anemia (hb < 8)
* Bone Marrow diseases
* Pregnancy and lactation
* Acute medical conditions/infections such as respiratory infections
* ventilatory support

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-01 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Functional Rating Scale - via questionnaire | 6 months

SECONDARY OUTCOMES:
Change in Appel Scale | 4 months
Change in SF-36 (The Short Form (36) Health Survey is a 36 Item) | 4 months
Change in Forced Vital Capacity (FVC) | 4 months

IPD SHARING:
Plan to Share IPD: Undecided